CLINICAL TRIAL: NCT00207584
Title: A Double-Blind, Randomized Placebo-Controlled Trial of Doxycycline for Chemoprophylaxis in the Setting of an Outbreak of Mycoplasma Pneumoniae
Brief Title: Randomized Controlled Trial of Doxycycline to Prevent Acquisition of Mycoplasma Pneumoniae in an Outbreak Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CDC-NCHSTP-9997
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Mycoplasma Pneumoniae

INTERVENTIONS:
Drug: Doxycycline treatment

SUMMARY:
This study was designed to determine whether taking daily doxycycline during an outbreak of Mycoplasma pneumoniae could prevent a person from getting infected and interrupt ongoing disease transmission during an outbreak. Doxycycline is a treatment for Mycoplasma pneumoniae, but it is not certain that the drug could prevent disease if used prophylactically.

ELIGIBILITY:
Inclusion Criteria:

- Working at hospital facility where outbreak of Mycoplasma pneumoniae occured

Exclusion Criteria:

- Pregnant, on antiseizure medications, allergic to macrolide antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1994-01; Study Completion 1994-04

CONTACTS AND LOCATIONS:
Overall Officials: Julia A Schillinger, MD, Principal Investigator — Centers for Disease Control and Prevention